CLINICAL TRIAL: NCT07176104
Title: Effects of Functional Bovine Milk Supplementation on Coronary In-Stent Restenosis and Major Adverse Cardiovascular Events in STEMI Patients Undergoing Primary PCI: A Randomized, Double-Blind, Controlled Trial
Brief Title: Functional Milk Supplementation to Reduce In-Stent Restenosis in STEMI Patients (SMASOEA Trial)
Acronym: SMASOEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raffaele Marfella (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor-Investigator, Raffaele Marfella, Professor, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMASOEA-STEMI-FM01
Record Dates: First submitted 2025-08-12; First posted 2025-09-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: ST-elevation Myocardial Infarction (STEMI); In-stent Restenosis
Keywords: ST-Elevation Myocardial Infarction; Inflammation
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Inflammation

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized, double-blind, controlled trial comparing functionalized milk versus non-functional milk in post-STEMI patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design. Participants, care providers, investigators, and outcomes assessors will be unaware of product allocation. Milk products will be packaged identically and coded by an independent pharmacist/dietary unit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Milk Group (Experimental): Participants will receive daily supplementation with functionalized bovine milk enriched with bioactive peptides and optimised lipid profile, in addition to guideline-directed secondary prevention therapy, for 12 months.
  Interventions: Dietary Supplement: Functional Bovine Milk
- Non-Functional Milk Group (Experimental): Participants will receive daily supplementation with an isocaloric non-functional bovine milk matched in appearance, taste, and packaging to the functionalized milk, in addition to guideline-directed secondary prevention therapy, for 12 months.
  Interventions: Dietary Supplement: Non-Functional Bovine Milk

INTERVENTIONS:
Dietary Supplement: Functional Bovine Milk — Functional milk product enriched with standardised bioactive peptides, provided daily for 12 months.
  Arms: Functional Milk Group
Dietary Supplement: Non-Functional Bovine Milk — Standard bovine milk with identical caloric and macronutrient profile to the functionalized milk, without enrichment, provided daily for 12 months.
  Arms: Non-Functional Milk Group

SUMMARY:
This randomized, double-blind, controlled clinical trial will evaluate the effects of daily supplementation with functionalized bovine milk, enriched with bioactive peptides and optimized lipid profile, on coronary in-stent restenosis and major adverse cardiovascular events (MACE) in patients with first ST-elevation myocardial infarction (STEMI) treated with primary percutaneous coronary intervention (PCI) and drug-eluting stent (DES) implantation. Participants will be randomly assigned to receive either functionalized milk or an isocaloric non-functional milk for 12 months, in addition to standard secondary prevention care. The primary endpoint is the incidence of in-stent restenosis at 12 months, assessed by coronary computed tomography angiography (CCTA). Secondary endpoints include MACE occurrence, metabolic and inflammatory biomarkers, oxidative stress markers, serum sirtuins, metabolomic profiles, and myocardial injury evaluated by cardiac positron emission tomography (PET). The study aims to determine whether functionalized milk can improve cardiovascular outcomes and modulate pathophysiological mechanisms after STEMI.

DETAILED DESCRIPTION:
Coronary artery disease remains a leading cause of morbidity and mortality worldwide. Despite advances in percutaneous coronary intervention (PCI) and the use of drug-eluting stents (DES), in-stent restenosis (ISR) continues to occur, driven by neointimal hyperplasia, vascular inflammation, and metabolic dysregulation. Nutritional interventions with specific bioactive compounds may offer an innovative adjunct to secondary prevention strategies.

This investigator-initiated, randomized, double-blind, controlled trial will assess whether functionalized bovine milk (FM) - standardized to contain a defined profile of bioactive peptides with antihypertensive, anti-thrombotic, anti-inflammatory, antioxidant, and plaque-stabilizing properties - can reduce ISR incidence and improve cardiovascular outcomes in patients with a first ST-elevation myocardial infarction (STEMI) treated with PCI and DES.

A total of 140 eligible patients will be randomized 1:1 to receive FM or an isocaloric non-functional milk (NFM) for 12 months, in addition to guideline-directed secondary prevention care. Both products will be organoleptically matched, blinded by coded packaging, and supplied in equal volumes.

The primary endpoint is the proportion of patients with ISR at 12 months, as measured by coronary computed tomography angiography (CCTA). Secondary endpoints include the composite of major adverse cardiovascular events (MACE: cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure), changes in insulin secretion and sensitivity, systemic inflammatory markers (hsCRP, IL-6, TNF-α), oxidative stress parameters, serum sirtuins, and metabolomic/lipidomic profiles obtained through LC-MS and GC-MS. Myocardial injury and viability will also be quantified by cardiac positron emission tomography (PET) at baseline and at study completion.

Adherence will be monitored through dietary records, packaging return counts, and optional biochemical markers. An independent Data Safety Monitoring Board (DSMB) will oversee patient safety and trial conduct. The study is powered to detect a 50% relative reduction in ISR (from 30% to 15%) with 80% power and a two-sided alpha of 0.05.

If positive, the trial will provide robust clinical evidence for the incorporation of a standardised functional dairy product into secondary prevention dietary guidelines for post-STEMI patients, potentially addressing both residual inflammatory risk and metabolic contributors to recurrent events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* First ST-elevation myocardial infarction (STEMI) treated with percutaneous coronary intervention (PCI) and drug-eluting stent implantation within the previous 4 weeks
* Stable clinical condition at enrollment
* Willingness to adhere to study procedures and dietary supplementation for 12 months
* Signed informed consent

Exclusion Criteria:

* Previous myocardial infarction or coronary revascularization
* Cardiogenic shock or severe heart failure (NYHA class IV)
* Severe renal impairment (eGFR <30 mL/min/1.73m²) or dialysis
* Active malignancy or life expectancy <1 year
* Known lactose intolerance or allergy to milk proteins
* Participation in another interventional clinical trial in the last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of In-Stent Restenosis at 12 Months | 12 months after PCI
  Proportion of patients presenting in-stent restenosis (ISR) as assessed by coronary computed tomography angiography (CCTA) at 12 months after index percutaneous coronary intervention (PCI) with drug-eluting stent.
Major Adverse Cardiovascular Events (MACE) | 12 months after PCI
  Composite endpoint of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, and hospitalization for heart failure.

SECONDARY OUTCOMES:
Change in Inflammatory Biomarkers | 12 months after PCI
  Change in hsCRP levels (mg/L)
Change in Oxidative Stress Parameters | 12 months after PCI
  Change from baseline in Change in plasma malondialdehyde (µmol/L).
Change in Serum Sirtuin Levels | 12 months after PCI
  Change from baseline in serum sirtuins as measured by ELISA.
Metabolomic Profile Changes | 12 months after PCI
  Variations in plasma metabolomic profiles assessed by LC-MS and GC-MS.
Cardiac PET Imaging Parameters | 12 months after PCI
  Change in myocardial perfusion and viability assessed by positron emission tomography.
Change in inflammatory markers | 12 months after PCIr PCI
  Change in IL-6 levels (pg/mL)
Change in inflammatory markers | 12 months after PCI
  Change in TNF-α levels (pg/mL)
Change in Oxidative Stress parameters | 12 months after PCI
  Change in 8-isoprostane levels (pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi della Campania "Luigi Vanvitelli" - Dipartimento di Scienze Mediche e Chirurgiche Avanzate, Napoli, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not yet been finalized. Data sharing will depend on ethical approval, participant consent, and compliance with applicable privacy regulations (including GDPR). If sharing is approved, anonymized datasets and related documentation may be made available to qualified researchers upon reasonable request, after publication of the primary results.

REFERENCES:
- [Result] Astrup A, Magkos F, Bier DM, Brenna JT, de Oliveira Otto MC, Hill JO, King JC, Mente A, Ordovas JM, Volek JS, Yusuf S, Krauss RM. Saturated Fats and Health: A Reassessment and Proposal for Food-Based Recommendations: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Aug 18;76(7):844-857. doi: 10.1016/j.jacc.2020.05.077. Epub 2020 Jun 17. PMID 32562735
- [Result] Lamarche B, et al. Dairy products and cardiovascular health: How strong is the evidence? J Am Coll Cardiol. 2016;67(12):1472-1489. doi:10.1016/j.jacc.2015.06.079. PMID: 27012404.
- [Result] Lordan R, Tsoupras A, Zabetakis I. Milk and dairy consumption: A review of cardiovascular health benefits and risks. Nutrients. 2018;10(8):993. doi:10.3390/nu10080993. PMID: 30087292.
- See also: Università degli Studi della Campania "Luigi Vanvitelli" — https://www.unicampania.it
- See also: Ministero dell'Agricoltura, della Sovranità Alimentare e delle Foreste (MASAF) — https://www.politicheagricole.it
- See also: National Institutes of Health — https://www.salute.it